CLINICAL TRIAL: NCT04696783
Title: Clinical Research on the Effect of PPI in Preventing Gastroesophageal Reflux Disease of Seafarers and Its Influence on Intestinal Flora and Mental State
Brief Title: The Effect of PPI in Preventing Gastroesophageal Reflux Disease of Seafarers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Li, The chief of the department of gastroenterology, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZDWY.XHNK.002
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Group (Experimental): Esomeprazole Magnesium Enteric-coated Tablets and lifestyle adjustment
  Interventions: Drug: Esomeprazole Magnesium Enteric-coated Tablets; Behavioral: Lifestyle adjustment
- non-Drug Group (Placebo Comparator): Only lifestyle adjustment
  Interventions: Behavioral: Lifestyle adjustment

INTERVENTIONS:
Drug: Esomeprazole Magnesium Enteric-coated Tablets — Nexium taken once every 2 days plus lifestyle adjustment
  Other Names: Nexium
  Arms: Drug Group
Behavioral: Lifestyle adjustment — Lifestyle adjustment

SUMMARY:
In view of the high incidence of GERD among seafarers and its continuing impact on the life quality of seafarers, it is necessary to use preventive treatment. At the same time, because both mental and psychological factors and changes in intestinal flora may play a certain role in the development and treatment of GERD, this project intends to take the seafarers involved in this scientific expedition as the participants to explore the effect of PPI discontinuous therapy in preventing gastroesophageal reflux disease of seafarers, a special occupational group and the changes in the mental and psychological status and intestinal flora of this group of people after PPI therapy.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the common digestive system diseases. However, at present, there are only sporadic reports on the diagnosis and treatment of seafarers' gastroesophageal reflux disease in the world, and there is a lack of systematic research and standardized diagnosis and treatment, especially in the prevention of GERD.

Seafarers work and live in a special marine environment for a long time and belong to a group of specific occupations. Studies have shown that the incidence of gastroesophageal reflux disease can be as high as 27% after 8 weeks of sailing, which is significantly higher than the prevalence of GERD worldwide. When single or multiple factors such as mental illness, high-fat diet, and changes in intestinal flora are combined, they have a significant additive effect and jointly promote the occurrence of GERD. In addition, the main treatment for gastroesophageal reflux disease is proton pump inhibitor (PPI), but long-term use of PPI may cause many adverse reactions. Because PPI can significantly increase the potential of hydrogen (PH) value in the stomach, long-term use of PPI to treat gastroesophageal reflux disease may cause changes in the microbiota colonized in the small and large intestines, and cause some symptoms related to intestinal flora disorders.

GERD is a chronic and recurrent disease that seriously affects the life quality. In addition to symptoms, gastroscopy and 24-hour esophageal pH testing are the main basis for diagnosis. However, during the voyage, the above procedures could not be carried out in time, resulting in delayed diagnosis and aggravated illness. Moreover, gastroscopy is generally suitable for people with alarm symptoms and it is not feasible for all people to receive gastroscopy,. In addition, although the 24-hour pH test is the gold standard for gastroesophageal reflux disease, it is generally used for people with negative gastroscopy and poor response to conventional treatment given the fact that it is invasive and there are not many hospitals that carry out the test. Because gastroesophageal reflux disease can be diagnosed clinically, in recent years, the gastroesophageal reflux disease questionnaire (Gerd Q) has been used for the preliminary clinical diagnosis of GERD. Studies have shown that with Gerd Q, family physicians and gastroenterologists have moderate or similar accuracy in the diagnosis of GERD. Many studies have shown that it has good authenticity and reliability. Therefore, this study did not use gastroscopy and 24-hour esophageal pH testing in the research steps, and the more practical Gerd Q scale was used for the diagnosis and evaluation of seafarers' GERD.

The first stage: record all seafarers'disease history/past history, demographic data, eating habits (whether there is high sugar, high fat, strong tea preference；whether drinking or smoking), vital signs, physical examination results, complete blood count, liver function, blood biochemistry, Gerd Q scale test and anxiety and depression scale evaluation, collect all seafarers' fecal samples before going to sea.

The second stage: After successful enrollment and intervention, the two groups of seafarers will be scored with Gerd Q and anxiety and depression scale every week, and fecal specimens of the two groups of seafarers will be collected for intestinal flora analysis. During the voyage, fecal specimens were collected in 5ml non-enzymatic drying tubes and stored in the -80℃ refrigerator on board. The entire intervention process continued until the end of the voyage.

The third stage: The efficacy evaluation stage.

ELIGIBILITY:
Inclusion Criteria:

* Agree to the implementation of this research and sign an informed consent form.

Exclusion Criteria:

* PPI drugs were previously used to treat acid-related diseases or conditions (including peptic ulcer, non-variceal upper gastrointestinal hemorrhage, gastroesophageal reflux disease, Zollinger-Ellison syndrome, and functional dyspepsia, eradication of Helicobacter pylori) 2 weeks before enrollment).
* Those having a history of stomach surgery.
* Those who have alarm symptoms (recent weight loss for unknown reasons, such as 5% or more of the original weight loss in the first half of the year; Progressive dysphagia, anemia, hematemesis, melena, hematochezia）or physical examination shows abnormalities such as abdominal rebound pain, masses, etc.).
* Pregnant or lactating women.
* Serious diseases and complications that may interfere with the research, such as heart, liver, kidney, lung, peripheral or autonomic nervous diseases, diabetes, etc.
* Allergic to PPI drugs.
* Having a history of drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Gerd Q score | 10 weeks
  The difference in the proportion of seafarers with a Gerd Q score of 8 or more between the two groups

SECONDARY OUTCOMES:
Anxiety and depression scores | 10 weeks
  Differences in anxiety and depression scores between the two groups
Intestinal flora analysis | 3 months
  Differences in intestinal flora in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shan, MD, Study Director — Fifth Affiliated Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
Individual participant data would not be available to other researchers in view of the confidentiality requirements of our research.